CLINICAL TRIAL: NCT00308035
Title: Foot Posture in People With Hemiplegia After Stroke
Brief Title: Foot Posture in People With Paralysis on One Side After Stroke
Status: Completed | Type: Observational
Sponsor: University of Kansas (Other)
Responsible Party: Patricia Kluding, PT PhD, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 10144
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
People who have had a stroke often have difficulty walking and problems with their balance. The purpose of this project is to examine problems with foot postures in people who have weakness on one side of their body

DETAILED DESCRIPTION:
The specific aims of this study are to:

1. Describe foot posture in individuals with hemiplegia following stroke using a quantitative navicular drop test.
2. Determine differences in people with normal, hypotonic, and hypertonic foot posture with regard to ankle range of motion, ankle strength, gait, and balance.

This is an observational design study to describe relationships between the variables. Measurements will include both descriptive and quantitative measures.

Thirty subjects with stroke will participate in one session of testing which will include: clinical assessment of foot posture using a descriptive classification system, quantitative measurement of navicular drop during standing, measurements of ankle range of motion, ankle strength, gait (lower extremity biomechanics and forceplate analysis), and static and dynamic balance. A chi-square test will be used to determine goodness of fit between classification with the descriptive system and the quantitative measurement. Independent one-way ANOVAs will be used to determine the mean differences in the foot posture groups for each of the dependent variables.

ELIGIBILITY:
Inclusion Criteria:

* subjects must have a diagnosis of a single stroke with resultant hemiplegia and be able to stand up from a seated position and walk 30 feet without assistance.

Exclusion Criteria:

* Subjects will be excluded if they present with significant foot or ankle pathology, other medical problem that would affect gait or balance, or language / cognitive deficits that would impair ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with hemiplegia from chronic stroke and limited ankle mobility
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2005-11; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kluding, PT PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States